

Research protocol

1 November 2017

**FINAL** version





# **Table of Contents**

| Protocol Details | 3 |
|----------------------------------------------------------------------|----|
| Signatures of all Investigators Involved in the Study | 4 |
| Summary | 5 |
| List of Abbreviations | 6 |
| List of Definitions | 7 |
| Background | 8 |
| Justification | 9 |
| Aim of Study | 9 |
| Investigation Plan | 10 |
| Study Population | 10 |
| Data | 11 |
| Statistical Analyses | 12 |
| Safety and Monitoring | 13 |
| Ethical Considerations | 13 |
| Conflict of Interest | 13 |
| Dissemination | 13 |
| References | 14 |
| Appendix 1: Penetrating Abdominal Trauma Index | |
| Appendix 2: Clavien-Dindo's Classification of Surgical Complications | 18 |
| Appendix 3: Surgical Site Infection defined by WHO | 19 |
| Appendix 4: Case Report Form | 20 |

#### Principal Investigator

Måns Muhrbeck, MD, Department of Surgery, Vrinnevi County Hospital, Linköping University, Norrköping, Sweden, e-mail: <a href="mans.muhrbeck@me.com">mans.muhrbeck@me.com</a>, mobile: +46-(0)70 333 88 52

#### Co-investigators

Andreas Älgå, MD, Centre for Research on Health Care in Disasters, Department of Public Health Sciences, Karolinska Institutet, Stockholm, Sweden; Rawand Musheer Haweizy, Lecturer, MBChB, MRCS, Emergency Hospital, Erbil, Iraq; Peter Andersson, MD, PhD, Associate Professor, Centre for Teaching and Research in Disaster Medicine and Traumatology, Linköping University, Linköping, Sweden; Andreas Wladis, MD, PhD, Professor, Centre for Teaching and Research in Disaster Medicine and Traumatology, Linköping University, Linköping, Sweden; Johan von Schreeb, MD, PhD, Associate Professor, Centre for Research on Health Care in Disasters, Department of Public Health Sciences, Karolinska Institutet, Stockholm, Sweden

#### **Protocol Details**

Version 1.9 Final 1 November 2017

# Signatures of all Investigators Involved in the Study

Måns Muhrbeck, MD<br/>Principal investigatorPeter Andersson, MD, PhD<br/>Co-investigatorRawand Musheer Haweizy, MD<br/>Co-investigatorJohan von Schreeb, MD, PhD<br/>Co-investigatorAndreas Wladis, MD, PhD<br/>Co-investigatorAndreas Älgå, MD<br/>Co-investigator

#### **Summary**

#### Study Rationale

The battle of Mosul was characterized by the use of improvised explosive devices, human shields and suicide bombers in an urban setting. It is unclear whether this type of warfare cause more extensive abdominal injuries to civilians than combatants. Understanding of the correlation between the severity of abdominal injuries, type of warfare and population affected is of importance when planning for surgical care in a conflict setting.

#### Aim

To assess whether civilians obtain more extensive abdominal injuries than combatants in an urban battle characterized by the use of indiscriminate weapons.

#### Study Design

An observational retrospective cohort study with longitudinal data collection.

All patients admitted with penetrating abdominal injury subjected to an exploratory laparotomy at Emergency Hospital, Erbil, between October 17, 2016 and July 16, 2017 will be included. Differences in demographics, injury mechanism, time since injury, clinical status on arrival, intraoperative findings, postoperative complications and outcome will be analysed.

#### Primary Objective

Differences in injury mechanism, organs injured, surgical treatment given, postoperative complications and outcome between civilians *and* combatants.

#### Secondary Objectives

Differences in surgical treatment given, postoperative complications and outcome between patients with prior surgical treatment of their injury *and* patients without prior surgical treatment.

Differences in surgical treatment given, postoperative complications and outcome between patients who receive surgical treatment less than 24 hours from injury *and* patients who receive surgical treatment more than 24 hours from injury will be analysed.

#### Statistical methods

Differences between groups will be analysed using t-test and regression models.

#### **List of Abbreviations**

EH Emergency Hospital, Erbil, Iraq

Ex-lap Exploratory laparotomy

ICRC International Committee of the Red Cross

IED Improvised Explosive Device

ISg Islamic State Group

WHO World Health Organization

#### **List of Definitions**

Civilians Children <16 years, all women and men ≥50

years.

Combatants Men 16-50 or combatants by own admission.

Exploratory laparotomy Surgical incision through the abdominal wall

into the abdominal cavity

PATI Penetrating Abdominal Trauma Index

Assess the severity of injury in patients with knife, gunshot or other penetrating wounds to

the abdomen (appendix 1).

Penetrating abdominal injury

An injury penetrating the peritoneum into the

abdominal cavity

Peritonitis Rigid involuntary general tenderness of the

abdominal wall.

Postoperative complication Any deviation from the ideal postoperative

course that is not inherent in the procedure and

does not comprise a failure to cure.

Classification of Surgical complications will be done according to Clavien-Dindo (appendix 2).

SSI Surgical Site Infection is present when one of

the following criteria are meet:

i. Purulent discharge from surgical site

ii. Positive culture

iii. Surgical site requires reopening

iv. SSI is present as judged by attending

physician

Severity according WHO guidelines

(appendix 3).

#### **Background**

#### Trail location

In 2014, Islamic State Group (ISg) made significant territorial gains in several governorates in Iraq and captured key cities, including Fallujah and Mosul<sup>1</sup>. ISg is unique among terrorist groups in that it employs a combination of conventional maneuverer warfare with tactics such as human shields, improvised explosive devices (IED's), suicide bombers and drones in order to capture and hold territory. These tactics are indiscriminate, leading to excessive civilian casualties<sup>2</sup>.

Emergency Hospital (EH) is one of two trauma hospitals in Erbil, a major metropolitan area in Kurdistan Region of Iraq. Erbil is located 94 kilometres east of the city of Mosul. Mosul is the provisional capital of the Nineveh region of Iraq. In mid-October 2016, the offensive to liberate Mosul from the ISg was initiated. EH was assigned by the Governate to exclusively provide care to injured from the armed conflict in and around Mosul. Since late December 2016 treatment facilities, run by other emergency care providers, have opened closer to Mosul. EH since then mainly served as a referral hospital.

The battle of Mosul formally ended on 10 July, 2017. The admission of causalities from Mosul to EH has since then diminished significantly. NGOs and other emergency care providers have also decreased their activities since.

Previous reports on exploratory laparotomy in conflict settings

Outcome of exploratory laparotomy (ex-lap) following war-related injuries has previously been extensively studied and reported on<sup>3-7</sup>. These reports have mainly concentrated on causes for and findings at ex-lap, and postoperative mortality (table 1). Few studies have focused on the differences in injury mechanism, complexity of injuries and outcome between civilians and combatants, especially in urban conflicts where IED's, human shields and suicide bombers are used<sup>2</sup>.

Table 1. Findings at ex-lap and postoperative mortality in different conflicts

| Conflict | Nb.<br>of<br>Ex-<br>laps | Negative explorations | Small<br>intestinal<br>injuries | Colon injuries incl. rectum | Other injuries | Postoperative mortality |
|---|---|---|---|---|---|---|
| Chad,1980 <sup>3</sup> | 210 | 4,8% | 33,0% | 21,1% | 32,7% | 22,5% |
| <b>Lebanon</b> 1975-85 <sup>4</sup> | 1314 | 9,7% | 24,7% | 21,2% | 55,0% | 9,5% |
| Former<br>Yugoslavia<br>1991-95 <sup>5</sup> | 93 | 4,3% | 30,0% | 28,4% | 41,5% | 10,8% |
| Gaza 2000-<br>03 <sup>6</sup> | 230 | 6,5% | 26,7% | 17,9% | 55,3% | 7,4% |
| Mosul,<br>Iraq, 2006 <sup>7</sup> | 153 | 15% | 23,7% | 18,7% | 57,6% | 33,3% |

#### **Justification**

There is a need for better understanding of demographics and outcome of ex-lap following abdominal injuries sustained in urban conflicts where IEDs, human shields and suicide bombers are used. The use of these indiscriminate weapons could affect civilians to a greater extent than combatants<sup>8</sup>. We therefore hypothesis that the use of indiscriminate weapons in an urban setting causes more extensive abdominal injuries to the civilian population than to combatants. The knowledge gained from this study could be crucial when planning surgical staffing and facility needs in similar contexts.

#### Potential Risks and Benefits

Since this is an observational retrospective cohort study without any interventional methods it poses little to no harm for the participants. A potential benefit for future patients would be an increase understanding among health care providers regarding what kind of abdominal injuries indiscriminate weapons causes. Furthermore, a better understanding on what impact the use of indiscriminate weapons have on the civilian population.

#### **Aim of Study**

To assess whether civilians have more complex abdominal injuries than combatants in an urban battle characterized by the use of indiscriminate weapons.

#### Primary Measure

Differences in injury mechanism, organs injured, surgical treatment given, postoperative complications and outcome between civilians *and* combatants.

#### Secondary Measures

Comparison of surgical treatment given, postoperative complications and outcome between patients with prior surgical treatment of their injury *and* patients without prior surgical treatment.

Differences in surgical treatment given, postoperative complications and outcome between patients who receive surgical treatment less than 24 hours from injury *and* patients who receive surgical treatment more than 24 hours from injury will be analysed.

See chapter Data, *patient files*, for detailed primary and secondary measurements.

#### **Investigation Plan**

Study Design

A cohort study with retrospective longitudinal data collection using routinely collected clinical data.

Study Period

Consecutive patients presenting at EH between October 17, 2016 and July 16, 2017 that meet eligibility criteria will be included. Patient history information preceding hospital admission will be included.

Study Location

Emergency Hospital, Erbil, Kurdistan Region, Iraq.

Study Duration for Participants

Participants will be followed from admission until discharged from EH.

#### **Study Population**

Recruitment Methods

Patients will be included from the surgical ledger at the Surgical Department of EH.

Inclusion Criteria

• All patients treated with ex-lap due to conflict-related penetrating injury presenting at EH between October 17, 2016 and July 31, 2017 will be included.

Exclusion Criteria

• Patients who received treatment several times during the study period will only be counted as one patient.

Information for Patients and Consent

Since this study is based on data from routine care participants will not be informed, nor will consent be asked of participation, as this could introduce bias and confounding factors. There are moreover no risks or potential gains involved for participants. No incentives or inducements will be provided to any participant or staff involved.

#### Data

#### Data Sources

Data was routinely prospectively collected on paper based patient forms in the clinical setting at EH. A *patient database* with consecutive patients treated between October 17, 2016 and July 31, 2017 was created. It is expected that the database will contain a total of 1,800 patients to produce approximately 160 evaluable subjects. Paper based *patient files* will be queried for demographic information, combatant or civilian status, admission dates, discharge dates, whether the injury was conflict-related or not, geographical site for injury, cause and mechanism of injury, prehospital data, medical history, vital signs at hospital admission, anatomical data and details regarding extent of abdominal injury, number and type of surgeries, details on surgery, need for ICU care, in hospital complications, re-admission including cause of re-admission, outcome including death and cause of death. Paper based data will be entered into a computer database using Epidata entry software (The Epidata Association, Odense, Denmark).

#### Patient Files

- Time of admission (specified)
- Age in years (specified)
- Sex (Male/Female/Unknown)
- Ethnicity (Arabic/Kurdish/Other/Unknown)
- Civilian/Combatant (Iraqi/Peshmerga/ISg/Unknown/Other)
- Time of injury (specified)
- Geographical location where injury occurred (specified)
- War-related injury (Yes/No/Unknown)
- Cause of injury (Bullet/Shell/Mie/IED/Unknown/Other)
- Mechanism of injury (Gunshot/Stab/Blast/Crush/Fragment/Burn/Traffic accident/Unknown/Other)
- Care prior to admission to EH (First Aid/Medical/Surgery/None given/Unknown)
- Provider of care prior to EH (MSF/Aspen/ICRC/Samaritan Purse/DoH/None)
- Mode of transport to EH (Military/Private car/Motorcycle/Ambulance/Unknown)
- Medical history (Healthy/Prior surgery/ Prior medical/Unknown)
- Body temperature (specified in Celsius)
- Heart rate (specified in beats/min)
- Blood pressure (specified in systole/diastole mmHg)
- Pregnant (Yes/No/Unknown)
- Pregnancy status based on (Lab/Question/Status/Unknown)
- Site and extent of abdominal wound (specified)
- Other injuries (Yes/No/Unknown, specified)
- Preoperative haemoglobin (specified in g/dL)
- Preoperative transfusions (Yes/No/Unknown, specified)
- Use of preoperative radiology (Yes/No/Unknown, specified)
- Time and date of procedure (specified)
- Duration of procedure (specified in hours and minute)

- Antibiotics prophylaxis (Yes/No/Unknown, specified)
- Procedure done (appendix 1 for definition of findings)
- Perioperative complication (Yes/No/Unknown, specified)
- Postoperative antibiotic prophylaxis (Yes/No/Unknown, specified)
- Postoperative infection (Yes/No/Unknown, appendix 3 for definition)
- Other postoperative complication (Yes/No/Unknown, appendix 2 for definition)
- Need of postoperative intensive care (Yes/No/Unknown, specified)
- Postoperative transfusions (Yes/No/Unknown, specified)
- Use of postoperative radiology (Yes/No/Unknown, specified)
- Further surgery done (Yes/No/Unknown, specified)
- Discharge (Yes/No/Unknown, specified)
- Follow-up scheduled (Yes/No/Unknown, specified)
- Re-admission (Yes/No/Unknown, specified)
- Deceased during hospital stay (Yes/No/Unknown, specified)
- Remarks

#### **Statistical Analyses**

#### Sample Size

Due to the nature of the study, the sample size will be a convenience sample of the available cases during the study period. It is expected that approximately 160 subjects will be enrolled.

#### Statistical Methods

Analysis will be done by as treated. A 5% significance level will be used. The difference in dichotomous, such as postoperative complication (primary outcome), and categorical outcomes with more than two categories will be tested using chi-square or Fisher test. For differences in continuous variables t-test will be used. In order to adjust our analysis for possible confounders and effect modifiers we will then use linear, logistic, ordinal or multinomial regression models, according to the nature of the outcome (continuous, binary, ordinal or nominal) with injury mechanism as the dependent variable and civilian/combatant as the main explanatory variable. Important demographic and injury specific parameters such as geographical location, date, age, sex, and injured organs, will then be included in the model as potential confounders.

#### Safety and Monitoring

#### Participant Confidentiality

The use of identification numbers will ensure anonymity in the data analysis. The participant's age, gender and demographic characteristics will be used as identifying features for analysis. The research team will ensure the ethical principles of beneficence, non-maleficence, justice and respect of patients are adhered to throughout the study.

#### Data Collection and Management

All data will remain anonymous throughout the data entry and analysis process. Nominal data will not be distributed outside the study location, or appear in any report or publication. Participant names will only be known by the research team. Identification codes will be safeguarded at EH facilities for the duration of the study.

#### **Ethical Considerations**

#### Ethics

The study will be conducted according to ethical principles stated in the Declaration of Helsinki<sup>9</sup>

#### Ethical Review Board Approval

An approval from the Ethics Review Committee of the Directorate of Health, Department of Health, Erbil, Kurdistan Regional Governate will be obtained before initiating the study.

#### **Conflict of Interest**

This is an investigator-initiated study. No company has had any influence over study design. There are no known conflicts of interest with other parties.

#### Dissemination

Printed and electronic versions of the final report will be provided to all partners involved in this research. Main findings will be presented orally to hospital staff at EH. The research methodology and results will be presented at scientific conferences and published in peer-reviewed journals.

#### References

- 1. Cockburn P. The rise of Islamic state: ISIS and the new Sunni revolution. London; New York: Verso 2015.
- 2. Affairs UNOfD. Improvised Explosive Devices (IEDs) [WWW]. New York, USA2016 [Available from: <a href="https://www.un.org/disarmament/convarms/ieds2/accessed 28 May 2017">https://www.un.org/disarmament/convarms/ieds2/accessed 28 May 2017</a>.
- 3. Dumurgier C WR, Durette D, Jancovici R, Suc L, Mechineau Y. Plaies de l'abdomen par projectiles de guerre: expérience du détachement médical de Kousseri- Riggil 15.07.80 au 15.12.80. [Abdominal wounds by the projectiles of war: experience of the medical detachment in Kousseri-Riggil 15.07.80 to 15.12.80.] Médecine et Hygiène 1992;40:2984-92.
- 4. Nassoura Z, Hajj H, Dajani O, et al. Trauma management in a war zone: the Lebanese war experience. The Journal of trauma 1991;31(12):1596-9.
- 5. Sikic N, Korac Z, Krajacic I, et al. War abdominal trauma: usefulness of Penetrating Abdominal Trauma Index, Injury Severity Score, and number of injured abdominal organs as predictive factors. Military medicine 2001;166(3):226-30.
- 6. Giannou C, Baldan M, Comité international de la Croix-Rouge. War surgery : working with limited resources in armed conflict and other situations of violence. Geneva: ICRC 2009.
- 7. Borhan MS A-NH. Analysis of Abdominal Missile Injuries: Prospective Study in Mosul., 2008.
- 8. Coupland RM, Samnegaard HO. Effect of type and transfer of conventional weapons on civilian injuries: retrospective analysis of prospective data from Red Cross hospitals. BMJ 1999;319(7207):410-2.
- 9. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA 2000;284(23):3043-5.
- 10. Moore EE, Dunn EL, Moore JB, et al. Penetrating abdominal trauma index. The Journal of trauma 1981;21(6):439-45.
- 11. Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg 2004;240(2):205-13.
- 12. Mentula PJ, Leppaniemi AK. Applicability of the Clavien-Dindo classification to emergency surgical procedures: a retrospective cohort study on 444 consecutive patients. Patient Saf Surg 2014;8:31. doi: 10.1186/1754-9493-8-31
- 13. Leaper DJ, Edmiston CE. World Health Organization: global guidelines for the prevention of surgical site infection. J Hosp Infect 2017;95(2):135-36. doi: 10.1016/j.jhin.2016.12.016

# **Appendix 1: Penetrating Abdominal Trauma Index**<sup>10</sup>

#### Overview

The Penetrating Abdominal Trauma Index (PATI) can be used to assess the severity of injury in patients with knife, gunshot or other penetrating wounds to the abdomen. The index can be used to compare performance of different emergency care settings.

#### Patient evaluation

- 1. 14 organs are examined
- 2. The risk associated with injury to each organ is graded from 1 to 5.
- 3. The estimated severity of each type of injury is graded from 1 to 5.

| Organ Injured | Risk<br>Factor | Injury | Injury<br>Estimate |
|---|---|---|---|
| Duodenum | 5 | single wall | 1 |
| | | ≤ 25% wall | 2 |
| | | >25% wall | 3 |
| | | duodenal wall and blood supply | 4 |
| | | pancreaticoduodenectomy | 5 |
| Pancreas | 5 | tangential | 1 |
| | | through-and-through (duct intact) | 2 |
| | | major debridement or distal duct injury | 3 |
| | | proximal duct injury | 4 |
| | | pancreaticoduodenectomy | 5 |
| Liver 4 | | nonbleeding peripheral | 1 |
| | | bleeding, central or minor debridement | 2 |
| | | major debridement or hepatic artery ligation | 3 |
| | | lobectomy | 4 |
| | | lobectomy with caval repair or extensive bilobar debridement | 5 |
| Large intestine | 4 | serosal | 1 |
| | | single wall | 2 |
| | | ≤ 25% wall | 3 |
| | | >25% wall | 4 |
| | | colon wall and blood supply | 5 |

| Major vascular | 4 | ≤ 25% wall | 1 |
|----------------|---|--------------------------------------|---|
| | | >25% wall | 2 |
| | | complete transection | 3 |
| | | interposition grafting or bypass | 4 |
| | | ligation | 5 |
| Spleen | 3 | nonbleeding | 1 |
| | | cautery or haemostatic agent | 2 |
| | | minor debridement or suturing | 3 |
| | | partial resection | 4 |
| | | splenectomy | 5 |
| Kidney | 3 | nonbleeding | 1 |
| | | minor debridement or suturing | 2 |
| | | major debridement | 3 |
| | | pedicle or major calyceal | 4 |
| | | nephrectomy | 5 |
| Extrahepatic 2 | | contusion | 1 |
| biliary | | cholecystectomy | 2 |
| | | ≤ 25% common duct wall | 3 |
| | | >25% common duct wall | 4 |
| | | biliary enteric reconstruction | 5 |
| Small bowel | 2 | single wall | 1 |
| | | through-and-through | 2 |
| | | ≤ 25% wall or 2-3 injuries | 3 |
| | | >25% wall or 4-5 injuries | 4 |
| | | wall and blood supply or >5 injuries | 5 |
| Stomach | 2 | single wall | 1 |
| | | through-and-through | 2 |
| | | minor debridement | 3 |
| | | wedge resection | 4 |
| | | >35% resection | 5 |
| Ureter | 2 | contusion | 1 |

| | laceration | 2 |
|---|---|---|
| | minor debridement | 3 |
| | segmental resection | 4 |
| | reconstruction | 5 |
| 1 | single wall | 1 |
| | through-and-through | 2 |
| | debridement | 3 |
| | wedge resection | 4 |
| | reconstruction | 5 |
| 1 | periosteum | 1 |
| | cortex | 2 |
| | through-and-through | 3 |
| | intra-articular | 4 |
| | major bone loss | 5 |
| 1 | nonbleeding small hematoma | 1 |
| | nonbleeding large hematoma | 2 |
| | suturing | 3 |
| | ligation of isolated vessels | 4 |
| | ligation of named vessels | 5 |
| | 1 | minor debridement segmental resection reconstruction 1 single wall through-and-through debridement wedge resection reconstruction 1 periosteum cortex through-and-through intra-articular major bone loss 1 nonbleeding small hematoma nonbleeding large hematoma suturing ligation of isolated vessels |

#### where:

• The percent injury to an organ wall probably indicates the portion of the entire circumference involved.

organ score = (risk factor)  $\times$  (injury estimate)

penetrating abdominal trauma index (PATI) = SUM (all injured organs)

#### Interpretation

minimum PATI: 0

• maximum PATI: 200

#### Risk of postoperative complications

- The risk of postoperative complications is low if the PATI is  $\leq 25$ .
- The rate of postoperative complications increases sharply if the PATI >25.

# **Appendix 2: Clavien-Dindo's Classification of Surgical Complications**<sup>11 12</sup>

| Grades | Definition |
|---|---|
| Grade I: | Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. |
| | Allowed therapeutic regimens are: drugs as antiemetic's, antipyretics, analgesic's, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside. |
| Grade II: | Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included. |
| Grade III: | Requiring surgical, endoscopic or radiological intervention |
| Grade III-a: | intervention not under general anaesthesia |
| Grade III-b: | intervention under general anaesthesia |
| Grade IV: | Life-threatening complication (including CNS complications) * requiring IC/ICU-management |
| Grade IV-a: | single organ dysfunction (including dialysis) |
| Grade IV-b: | multi organ dysfunction |
| Grade V: | Death of a patient |
| Suffix 'd': | If the patients suffers from a complication at the time of discharge, the suffix "d" (for 'disability') is added to the respective grade of complication. This label indicates the need for a follow-up to fully evaluate the complication. |

<sup>‡</sup> brain haemorrhage, ischemic stroke, subarachnoidal bleeding, but excluding transient ischemic attacks (TIA); IC: Intermediate care; ICU: Intensive care unit.

# Appendix 3: Surgical Site Infection defined by WHO<sup>13</sup>

- Superficial incisional, affecting the skin and subcutaneous tissue. These infections may be indicated by localized signs such as redness, pain, heat or swelling at the site of the incision or by the drainage of pus.
- Deep incisional, affecting the fascial and muscle layers. These infections may be indicated by the presence of pus or an abscess, fever with tenderness of the wound, or a separation of the edges of the incision exposing the deeper tissues.
- Organ or space infection, which involves any part of the anatomy other than the
  incision that is opened or manipulated during the surgical procedure, for example
  joint or peritoneum. These infections may be indicated by the drainage of pus or
  the formation of an abscess detected by histopathological or radiological
  examination or during re-operation. Organ infection is not included within the
  scope of this guideline.

## **Appendix 4: Case Report From**



# Exploratory laparotomy following penetrating abdominal injuries: a cohort study from a referral hospital in Erbil, Kurdistan region in Iraq

**Case Report Form** 

1 November 2017

**FINAL version** 





Case Report From (CRF), version 171101, protocol:

| レコ | ıΤı | $\triangle$ | n | Τ. | ۱ ۱ | 12 | ナコ |
|----|-----|-------------|---|----|-----|----|----|
| Pa | ıuı | $\Box$ | ш | L | U | a | ιa |

| Patient no | | | | |
|---|---|---|---|---|
| 1. Time of admission | day month | year | : hours minutes | Unknown |
| 2. Age | | in years | Unknown | |
| 3. Sex | Male | Female | Unknown | |
| 4. Ethnicity | Arabic | Kurdish | Other | Unknown |
| If other, specify | | | | |
| 5. Civilian/Combatant | Civilian | Combatant | Unknown | |
| If combatant | Iraqi Unknown | Peshmerga Other | IS | |
| If other, specify | | | | |
| Investigators signature | | | / /<br>day month | year |







| Case Report From (CRF), vers | sion 171101, protocol | : | |
|---|---|---|---|
| Injury Data | | | |
| Patient no | | | |
| 6. Time of injury | : | / / | II.I. |
| | hours minutes | day month year | Unknowr |
| 7. Geographical location wh | ere injury occurred | | |
| Al Uraybi Ar Rafat L Ar Rabi Al Islah As Sinaa al-Zerai Abu Tammam Al Yarmuk | Al Musarit Shurta Ah Muthanna Ath haqafah As S | Al Cahira Az Zuhoor Al Bakir An Nur Sihhah Arbajiyah Al Kadra Al Quds Al Intisar Al Wahda Al Intisar O 1 2 3 k | n. |
| | | Unknown Other | |
| If other, specify location where inju | ury occurred | | |
| Investigators signature | | day month ye | ar |



| Case Report From (CRF), version 1 | 71101, pro | tocol: | |
|---|---|---|---|
| Injury Data continued | | | |
| Patient no | | | |
| 8. War-related injury | Yes | No | Unknown |
| 9. Cause of injury (If several causes number in same order as question 20 and 21) | Bullet IED | Shell Unknown | Mine Other |
| If other, specify | | | |
| 10. Mechanism of injury (If several number in same order as question 20 and 21) | Gunshot Crush Burn | Stab Fragment Other | Blast Unknown Traffic accident |
| If other, specify | | | |
| Investigators signature | | | / /<br>day month year |



Exploratory laparotomy following penetrating abdominal injuries: a cohort study from a referral hospital in Erbil, Kurdistan region in Iraq Case Report From (CRF), version 171101, protocol: Prehospital Care Data Patient no

| 11. Care prior to admission to EH (If several number in chronological order) | First aid Unknown | Medical Surgery | None given |
|---|---|---|---|
| If surgery, specify procedure done | | | |
| | / day month | | rocedure |
| <b>12. Provider of care prior to EH</b> (If several number in chronological order) | MSF | Aspen | ICRC |
| | Unknown | Samaritan Pur | rse |
| | None | Department o | f Health |
| Other, specify | | | |
| Investigators signature | | | / / |

day



month



Exploratory laparotomy following penetrating abdominal injuries: a cohort study from a referral hospital in Erbil, Kurdistan region in Iraq Case Report From (CRF), version 171101, protocol: Prehospital Care Data cont. Patient no 13. Mode of transport to EH (If several number in chronological order) Military Private car Motorcycle Ambulance Unknown Other, specify 14. Medical history Healthy Unknown Prior surgery Prior medical If prior surgery specify procedure(s) If prior medical condition(s) specify Investigators signature day month







| Case Report From (CRF), version 171 | 101, protocol: _ | | | |
|---|---|---|---|---|
| Clinical Data at OPD | | | | |
| Patient no | | | ] | |
| 15. Body temperature | | in Celsius. | Unkr | nown |
| 16. Heart rate | | in beats/min | Unkr | nown |
| 17. Blood pressure | /<br>Systole | in mmI<br>Diastole | Hg Unkr | nown |
| 18. Pregnant | Yes | No | Unknown | |
| 19. Pregnancy status based on | Lab | Question | Status | Unknown |
| 20. Site and extent of abdominal wo | ound | | | |
| 11:11 | 1 | | 1 | If >2 injuries use remarks |
| Mark each wound by number | | | | |
| 1. | | | | |
| Brief description of size and depth | | | | |
| 2. | | | | |
| Brief description of size and depth | | | | |
| Investigators signature | | | day mont | th year |

| ol: |
|-----|
|-----|

### Clinical Data at OPD cont.

#### Patient no

### 21. Other injuries





If >3 injuries use remarks

Karolinska Institutet

Mark each wound by number

| 1. | | | |
|-------------------------------------|-----|-------|------|
| Brief description of size and depth | | | |
| 2. | | | |
| Brief description of size and depth | | | |
| 3. | | | |
| Brief description of size and depth | | | |
| Investigators signature | / | / | |
| | day | month | year |
| | | | _ |

Case Report From (CRF), version 171101, protocol: Preoperative Data Patient no g/dL 22. Preoperative haemoglobin Unknown 23. Preoperative transfusions None given Unknown Units of whole blood Units of packed red blood cells Units of Platelets Units of Plasma 24. Use of preoperative radiology No Unknown Computed Tomography (CT) If CT was used, specify findings Conventional radiology (X-ray) If X-ray was used, specify findings Investigators signature



day

month

year



# Case Report From (CRF), version 171101, protocol: Operative Data Patient no 25. Time and date of procedure hours minutes day month Unknown year 26. Duration of procedure hours minutes Unknown 27. Antibiotics prophylaxis No Yes Unknown If yes, specify type, dose and duration 28. Procedure done If lack of space use remarks (If several procedures are relevant. Mark most relevant with S.) Primary haemostasis (damage control) Yes No Unknown Removal of foreign bodies Yes No Unknown Raphi of bowel No Yes Unknown If raphi, specify site(s) and count(s) Small intestinal resection with anastomosis Yes No Unknown If anastomosis, specify site(s) and technique(s) Investigators signature





| Case Report From (CRF), version 171101, | , protocol: | | |
|---|---|---|---|
| Operative Data cont. Patient no | | | |
| <b>Procedure done cont.</b> Colon resection with anastomosis | Yes | No | Unknown |
| If anastomosis, specify site(s) and technique(s) | | | |
| Stoma/Bowel deviation | Yes | No | Unknown |
| If stoma(s), specify site(s) and technique(s) | | | |
| Vascular repair | Yes | No | Unknown |
| If vascular repair(s), specify location(s) and techn | ique(s) | | |
| Splenectomy | Yes | No | Unknown |
| Other | Yes | No | Unknown |
| If other(s), specify location(s) and procedure(s) | | | |
| 29. Perioperative complication | Yes | No | Unknown |
| If yes, specify type | | | |
| Investigators signature | | | / / day month year |
| Validated by and date: | E | Emergency Managmen<br>ری جاره سه ری فرباگورای | t Center of the state of the st |

Exploratory laparotomy following penetrating abdominal injuries: a cohort study from a referral hospital in Erbil, Kurdistan region in Iraq Case Report From (CRF), version 171101, protocol:

| Postoperative Data | |
|---|---|
| Patient no | |
| <b>30. Postoperative antibiotic prophylaxis</b> (without treating a defined infection) | No Unknown Yes |
| If yes, specify type, doses and duration | |
| 31. Postoperative infection (If several is possible mark all with with appropriate postop. day.) | No Unknown Appendix 3 for definition |
| Affecting the skin and subcutaneous tissue | / / Date of diagnosis day month year |
| Affecting the fascial and muscle layers | / / Date of diagnosis |
| Affecting abdominal cavity | / / Date of diagnosis |
| Sepsis | / / Date of diagnosis |
| Measures taken (for ex. intensive care, iv antibiotics | s, dialysis) |
| Unspecified infection | / / Date fo diagnosis |
| Explain and measures taken | |
| Investigators signature | |







| Case Report From (CRF), version 171101, p | protocol: |
|---|---|
| Postoperative Data cont. Patient no | |
| 32. Other postoperative complication | No Unknown Appendix 2 for definiton |
| Yes | / / Date of diagnosis day month year |
| Type and measures taken | |
| 33. Need of postoperative intensive care | No Unknown Yes |
| If yes, specify reason(s) for intensive care | |
| Discharged from Intensive Care Unit | / / Date |
| 34. Postoperative transfusions | None given Unknown |
| | Units of whole blood |
| | Units of packed red blood cells |
| | Units of Platelets |
| | Units of Plasma |
| 35. Use of postoperative radiology | No Unknown CT X-ray |
| If use of radiology, specify findings | |
| Investigators signature | |
| Validated by and date: | Emergency Managment Center المعالمة ال |

Exploratory laparotomy following penetrating abdominal injuries: a cohort study from a referral hospital in Erbil, Kurdistan region in Iraq Case Report From (CRF), version 171101, protocol: Postoperative Data cont. Patient no 36. Further surgery done Date No Unknown 1.Yes If yes, specify procedure done Date 2.Yes If yes, specify procedure done Date 3.Yes If yes, specify procedure done Investigators signature



Exploratory laparotomy following penetrating abdominal injuries: a cohort study from a referral hospital in Erbil, Kurdistan region in Iraq Case Report From (CRF), version 171101, protocol: Postoperative Data cont. Patient no 37. Discharge No Unknown Date of discharge day month year **Discharged Status** Hospital care complete Left Against Medical Advice Unknown Transferred for further care Transferred to where Type of care planned Investigators signature day month



Exploratory laparotomy following penetrating abdominal injuries: a cohort study from a referral hospital in Erbil, Kurdistan region in Iraq Case Report From (CRF), version 171101, protocol: Postoperative Data cont. Patient no 38. Follow-up scheduled No Yes Unknown When and reason for follow-up 39. Re-admission No Yes Unknown Date of re-admission day month year Reason for re-admission 40. Deceased during hospital stay No Yes Unknown Cause of death Unknown Date of death day month year

| Emergency Management Center و المراجعة | LINKÖPING UNIVERSITY |
|---|---|
| | EMC Emergency Management Center من المسلم ا |

day

month

year

Investigators signature

| Exploratory laparotomy following penetrating abdom Erbil, Kurdistan region in Iraq | ninal injuries: a cohort study from a re | ferral ho | ospital in | |
|---|---|---|---|---|
| Case Report From (CRF), version 171101, p | protocol: | | | |
| Postoperative Data cont. | | | | |
| Patient no | | | | |
| 41. Remarks | | | | |
| Investigators signature | | / | / | |
| | | day | month | year |

